CLINICAL TRIAL: NCT00931606
Title: A Phase 2, Double-blind, Randomized, Placebo-Controlled Study of ACE-011 for the Treatment of Chemotherapy Induced Anemia in Patients With Metastatic Breast Cancer
Brief Title: Study of Sotatercept for the Treatment of Chemotherapy Induced Anemia in Patients With Metastatic Breast Cancer (MK-7962-012)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: administrative reasons (slow patient enrollment)
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7962-012; A011-08 (Other: Acceleron pharma); MK-7962-012 (Other: Merck)
Record Dates: First submitted 2009-05-22; First posted 2009-07-02 (Estimated); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Chemotherapy Induced Anemia
Keywords: anemia; metastatic; breast; cancer
MeSH Terms: conditions — Anemia; Neoplasm Metastasis; Neoplasms | interventions — ACE-011

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sotatercept 0.1 mg/kg (Experimental): Participants will receive sotatercept 0.1 mg/kg subcutaneously every 28 days up to 4 doses.
  Interventions: Biological: Sotatercept
- Sotatercept 0.3 mg/kg (Experimental): Participants will receive sotatercept 0.3 mg/kg subcutaneously every 28 days up to 4 doses.
  Interventions: Biological: Sotatercept
- Sotatercept 0.5 mg/kg (Experimental): Participants will receive sotatercept 0.5 mg/kg subcutaneously every 28 days up to 4 doses.
  Interventions: Biological: Sotatercept
- Placebo (Placebo Comparator): Participants will receive placebo subcutaneously every 28 days up to 4 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Sotatercept — up to 4 subcutaneous doses of sotatercept given once every 28 days
  Other Names: ACE-011
  Arms: Sotatercept 0.1 mg/kg; Sotatercept 0.3 mg/kg; Sotatercept 0.5 mg/kg
Drug: Placebo — up to 4 subcutaneous doses of placebo given once every 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the percentage of participants in each sotatercept dose regimen who achieve a hematopoietic response during the treatment period including up to 2 months after the last dose of sotatercept treatment of chemotherapy-induced anemia (CIA) in participants with metastatic breast cancer. Hematopoietic response was defined as an increase in hemoglobin concentration of ≥ 1 g/dL relative to baseline for 28 consecutive days during the treatment period including up to 2 months after the last dose of sotatercept in the absence of red blood cell (RBC) transfusion or treatment with an erythropoiesis-stimulating agent (ESA).

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed diagnosis of breast cancer documented by cytology or biopsy.
* Has evidence of metastatic breast cancer with a minimum of one lesion per Response Evaluation Criteria in Solid Tumors v 1.1 (RECIST v 1.1) criteria.
* Is receiving a chemotherapy regimen including one of the following: anthracycline, taxane, gemcitabine, vinorelbine or capecitabine.
* Has planned treatment with the same chemotherapy regimen for a minimum of 9 weeks after Day 1 of study intervention administration.
* ≥ 30 days elapsed (from Day 1) since previous treatment with an erythropoiesis stimulating agent (ESA) (including treatment with intravenous (IV) iron) for chemotherapy induced anemia.
* ≥ 7 days elapsed (from Day 1) since the last red blood cell (RBC) transfusion and receipt of ≤ 2 units of blood in the past 30 days.
* Life expectancy of ≥ 6 months.

Exclusion Criteria:

* Has had prior radiation therapy to > 20% of the whole skeleton.
* Has had > 5 prior chemotherapy treatment regimens for metastatic breast cancer.
* Has a history of autoimmune or hereditary hemolysis or gastrointestinal bleeding.
* Has clinically significant pulmonary, endocrine, neurologic, gastrointestinal, hepatic or genitourinary disease unrelated to underlying hematologic disorder.
* Has heart failure as classified by the New York Heart Association (NYHA) classification of 3 or higher.
* Has a recent history of thrombosis, deep vein thrombosis (DVT), pulmonary emboli, or embolic stroke, occurring within the last 6 months.
* Has untreated central nervous system (CNS) metastases or CNS metastases treated with whole brain radiotherapy < 6 months prior to Day 1.
* Has a diagnosis of a myeloid malignancy or known history of myelodysplasia.
* Has a history of second malignancy within 5 years (except excised and cured basal cell carcinoma, squamous cell carcinoma of the skin or cervical carcinoma in situ).
* Has had administration of IV antibiotics or febrile (temperature elevation > 38 ° C) within 14 days of Day 1.
* Has uncontrolled hypertension.
* Has known history of hepatitis B surface antigen (HBsAg and HB core antibody (Ab)), human immunodeficiency virus (HIV) antibody or active hepatitis C.
* Has clinically significant iron (transferrin saturation < 20%), vitamin B12, or folate deficiency.
* Has a history of anemia as a result of inherited hemoglobinopathy such as sickle cell anemia or thalassemia.
* Has a history of autoimmune or hereditary hemolysis; active gastrointestinal bleeding (within the last 6 months as compared to Day 1).
* Has received treatment with another investigational drug or device within 1 month prior to Day 1.
* Is pregnant or lactating.
* Has a history of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational product.
* Has had major surgery within 30 days prior to Day 1 (patients must have completely recovered from any previous surgery prior to Day 1).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2010-11-18 (Actual); Study Completion 2010-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp and Dohme LLC
Locations (35):
- United States (28):
  - Investigative Site, Sedona, Arizona
  - Investigative Site, Hot Springs, Arkansas
  - Investigative Site, Beverly Hills, California
  - Investigative Site, Corona, California
  - Investigative Site, Fountain Valley, California
  - Investigative Site, Montebello, California
  - Investigative Site, Riverside, California
  - Investigative Site, Denver, Colorado
  - Investigative Site, Boynton Beach, Florida
  - Investigative Site, Hinsdale, Illinois
  - Investigative Site, Evansville, Indiana
  - Investigative Site, Wichita, Kansas
  - Investigative Site, Baltimore, Maryland
  - Investigative Site, Grand Rapids, Michigan
  - Investigative Site, Tupelo, Mississippi
  - Investigative Site, Kansas City, Missouri
  - Investigative Site, Nyack, New York
  - Investigative Site, Goldsboro, North Carolina
  - Investigative Site, High Point, North Carolina
  - Investigative Site, Winston-Salem, North Carolina
  - Investigative Site, Bismarck, North Dakota
  - Investigative Site, Middletown, Ohio
  - Investigative Site, Philadelphia, Pennsylvania
  - Investigative Site, Charleston, South Carolina
  - Investigative Site, Austin, Texas
  - Investigative Site, Dallas, Texas
  - Investigative Site, Tyler, Texas
  - Investigative Site, Lacey, Washington
- Russia (7):
  - Investigative Site, Krasnodar
  - Investigative Site, Moscow
  - Investigative Site, Nizhny Novgorod
  - Investigative Site, Nizhny Novograd (2)
  - Investigative Site, Pyatigorsk
  - Investigative Site, Saint Petersburg
  - Investigative Site, Stavropol

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Raftopoulos H, Laadem A, Hesketh PJ, Goldschmidt J, Gabrail N, Osborne C, Ali M, Sherman ML, Wang D, Glaspy JA, Puccio-Pick M, Zou J, Crawford J. Sotatercept (ACE-011) for the treatment of chemotherapy-induced anemia in patients with metastatic breast cancer or advanced or metastatic solid tumors treated with platinum-based chemotherapeutic regimens: results from two phase 2 studies. Support Care Cancer. 2016 Apr;24(4):1517-25. doi: 10.1007/s00520-015-2929-9. Epub 2015 Sep 14. PMID 26370220
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was terminated early after 30 participants were enrolled due to slower than expected rate of enrollment as a result of changes in guidance for the treatment of participants with breast cancer and chemotherapy induced anemia (CIA).
Groups:
- Sotatercept 0.1 mg/kg: Participants received sotatercept 0.1 mg/kg subcutaneously every 28 days up to 4 doses.
- Sotatercept 0.3 mg/kg: Participants received sotatercept 0.3 mg/kg subcutaneously every 28 days up to 4 doses.
- Sotatercept 0.5 mg/kg: Participants received sotatercept 0.5 mg/kg subcutaneously every 28 days up to 4 doses.
- Placebo: Participants received placebo subcutaneously every 28 days up to 4 doses.
Period: Overall Study
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Started | 8 | 10 | 7 | 5
Completed | 3 | 1 | 1 | 2
Not Completed | 5 | 9 | 6 | 3
Not completed — Death | 1 | 3 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 3 | 0
Not completed — Sponsor Decision | 1 | 4 | 0 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo | Total
Number analyzed (Participants) | 8 | 10 | 7 | 5 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.6 (9.38) | 50.8 (8.51) | 55.6 (12.53) | 49.2 (10.62) | 51.9 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 7 | 5 | 30
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 8 | 10 | 7 | 4 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: Kilograms] — Participants weight in kilograms is presented as the mean for each treatment arm.
  Kilograms | 67.38 (18.338) | 71.80 (9.500) | 69.94 (9.953) | 79.62 (9.926) | 71.49 (12.647)
Chemotherapy Frequency [Count of Participants; unit: Participants] — Chemotherapy frequency among the Modified Intent to Treat Group was differentiated as either weekly or less frequently for participants.
  Participants
    Weekly | 2 | 2 | 1 | 1 | 6
    Less Frequently | 6 | 8 | 6 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Hematopoietic Response
Description: Hematopoietic response rate is defined as the percentage of participants who had increase in hemoglobin concentration of ≥ 1 g/dL relative to baseline for 28 consecutive days during the treatment period including up to 2 months after the last dose of study treatment in the absence of red blood cell (RBC) transfusion or treatment with an erythropoiesis-stimulating agent (ESA). The percentage of participants who achieved hematopoietic response is presented.
Time Frame: Baseline and Up to ~145 Days
Population: All randomized participants who have confirmed CIA, received at least one dose of study intervention and on study intervention for at least 2 months (57 days).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- All Sotatercept-treated Participants: Participants received sotatercept at one of the following doses: 0.1 mg/kg, 0.3 mg/kg, or 0.5 mg/kg subcutaneously every 28 days up to 4 doses.
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo | All Sotatercept-treated Participants
Number analyzed (Participants) | 5 | 9 | 4 | 5 | 18
Percentage of Participants
  Overall | 0 [0 to 52.2] | 33.3 [7.5 to 70.1] | 50.0 [6.8 to 93.2] | 20.0 [0.5 to 71.6] | 27.8 [9.7 to 53.5]
  Received weekly chemotherapy and showed a response: number analyzed (Participants) | 2 | 2 | 1 | 1 | 5
  Received weekly chemotherapy and showed a response | 0 [0 to 84.2] | 0 [0 to 84.2] | 25.0 [2.5 to 100.0] | 20 [2.5 to 100.0] | 5.6 [0.5 to 71.6]
  Received less frequent chemotherapy and showed a response: number analyzed (Participants) | 3 | 7 | 3 | 4 | 13
  Received less frequent chemotherapy and showed a response | 0 [0 to 70.8] | 33.3 [9.9 to 81.6] | 25.0 [0.8 to 90.6] | 0 [0 to 60.2] | 22.2 [9.1 to 61.4]
Statistical Analysis 1: Comparison: Sotatercept 0.1 mg/kg vs Placebo; Overall; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 2: Comparison: Sotatercept 0.3 mg/kg vs Placebo; Overall; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 3: Comparison: Sotatercept 0.5 mg/kg vs Placebo; Overall; Test type: Superiority; p = 0.524, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 4: Comparison: Placebo vs All Sotatercept-treated Participants; Overall; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 5: Comparison: Sotatercept 0.1 mg/kg vs Placebo; Weekly Chemotherapy; Test type: Superiority; p = 0.333, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 6: Comparison: Sotatercept 0.3 mg/kg vs Placebo; Weekly Chemotherapy; Test type: Superiority; p = 0.333, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 7: Comparison: Placebo vs All Sotatercept-treated Participants; Weekly Chemotherapy; Test type: Superiority; p = 0.333, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 8: Comparison: Sotatercept 0.3 mg/kg vs Placebo; Less Frequent Chemotherapy; Test type: Superiority; p = 0.236, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 9: Comparison: Sotatercept 0.5 mg/kg vs Placebo; Less Frequent Chemotherapy; Test type: Superiority; p = 0.429, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 10: Comparison: Placebo vs All Sotatercept-treated Participants; Less Frequent Chemotherapy; Test type: Superiority; p = 0.519, Fisher Exact; Clopper and Pearson exact approach

2. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experienced AEs is reported.
Time Frame: Up to ~175 Days
Population: All participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 8 | 10 | 7 | 5
Participants | 6 | 7 | 7 | 5

3. Secondary Outcome: Number of Participants Who Discontinued Study Intervention Due to an Adverse Event
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants discontinuing study intervention due to AEs is reported.
Time Frame: Up to ~85 Days
Population: All participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 8 | 10 | 7 | 5
Participants | 1 | 0 | 4 | 1

4. Secondary Outcome: Percentage of Participants Achieving an Increase From Baseline Hemoglobin of ≥ 2 g/dL
Description: Percentage of participants achieving an increase from baseline hemoglobin of ≥ 2 g/dL for 28 consecutive days during the treatment period and up to 2 months after the last dose of study treatment in the absence of RBC transfusion or treatment with an ESA. The percentage of participants achieving an increase from baseline hemoglobin of ≥ 2 g/dL for 28 consecutive days is presented.
Time Frame: Baseline and Up to ~145 Days
Population: All randomized participants who have confirmed CIA, received at least one dose of study intervention and on study treatment for at least 2 months (57 days).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo | All Sotatercept-treated Participants
Number analyzed (Participants) | 5 | 9 | 4 | 5 | 18
Percentage of Participants
  Overall | 0 [0 to 52.2] | 11.1 [0.3 to 48.2] | 0 [0 to 60.2] | 0 [0 to 52.2] | 5.6 [0.1 to 27.3]
  Received weekly chemotherapy and showed a response: number analyzed (Participants) | 2 | 2 | 1 | 1 | 5
  Received weekly chemotherapy and showed a response | 0 [0 to 84.2] | 0 [0 to 84.2] | 0 [0 to 97.5] | 0 [0 to 97.5] | 0 [0 to 52.2]
  Received less frequent chemotherapy and showed a response: number analyzed (Participants) | 3 | 7 | 3 | 4 | 13
  Received less frequent chemotherapy and showed a response | 0 [0 to 70.8] | 11.1 [0.4 to 57.9] | 0 [0 to 70.8] | 0 [0 to 60.2] | 5.6 [0.2 to 36.0]
Statistical Analysis 1: Comparison: Sotatercept 0.3 mg/kg vs Placebo; Overall; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 2: Comparison: Placebo vs All Sotatercept-treated Participants; Overall; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 3: Comparison: Sotatercept 0.3 mg/kg vs Placebo; Less Frequent Chemotherapy; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 4: Comparison: Placebo vs All Sotatercept-treated Participants; Less Frequent Chemotherapy; Test type: Superiority; p > 0.999, Fisher Exact; Clopper and Pearson exact approach

5. Secondary Outcome: Percentage of Participants Achieving an Increase From Baseline Hemoglobin ≥ 11 g/dL
Description: Percentage of participants achieving hemoglobin ≥ 11 g/dL for 28 consecutive days during the treatment period and up to 2 months after the last dose of study treatment in the absence of RBC transfusion or treatment with an ESA. The percentage of participants achieving an increase from baseline hemoglobin of ≥ 11 g/dL for 28 consecutive days is presented.
Time Frame: Baseline and Up to ~145 Days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo | All Sotatercept-treated Participants
Number analyzed (Participants) | 5 | 9 | 4 | 5 | 18
Percentage of Participants
  Overall | 20.0 [0.5 to 71.6] | 22.2 [2.8 to 60.0] | 75.0 [19.4 to 99.4] | 20.0 [0.5 to 71.6] | 33.3 [13.3 to 59.0]
  Received weekly chemotherapy and showed a response: number analyzed (Participants) | 2 | 2 | 1 | 1 | 5
  Received weekly chemotherapy and showed a response | 0 [0 to 84.2] | 11.1 [1.3 to 98.7] | 25.0 [2.5 to 100.0] | 20.0 [2.5 to 100.0] | 11.1 [5.3 to 85.3]
  Received less frequent chemotherapy and showed a response: number analyzed (Participants) | 3 | 7 | 3 | 4 | 13
  Received less frequent chemotherapy and showed a response | 20.0 [0.8 to 90.6] | 11.1 [0.4 to 57.9] | 50.0 [9.4 to 99.2] | 0 [0 to 60.2] | 22.2 [9.1 to 61.4]
Statistical Analysis 1: Comparison: Sotatercept 0.1 mg/kg vs Placebo; Overall; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999, are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 2: Comparison: Sotatercept 0.3 mg/kg vs Placebo; Overall; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 3: Comparison: Sotatercept 0.5 mg/kg vs Placebo; Overall; Test type: Superiority; p = 0.206, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 4: Comparison: Placebo vs All Sotatercept-treated Participants; Overall; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 5: Comparison: Sotatercept 0.1 mg/kg vs Placebo; Weekly Chemotherapy; Test type: Superiority; p = 0.333, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 6: Comparison: Sotatercept 0.3 mg/kg vs Placebo; Weekly Chemotherapy; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999, are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 7: Comparison: Placebo vs All Sotatercept-treated Participants; Weekly Chemotherapy; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999, are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 8: Comparison: Sotatercept 0.1 mg/kg vs Placebo; Less Frequent Chemotherapy; Test type: Superiority; p = 0.429, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 9: Comparison: Sotatercept 0.3 mg/kg vs Placebo; Less Frequent Chemotherapy; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 10: Comparison: Sotatercept 0.5 mg/kg vs Placebo; Less Frequent Chemotherapy; Test type: Superiority; p = 0.143, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 11: Comparison: Placebo vs All Sotatercept-treated Participants; Less Frequent Chemotherapy; Test type: Superiority; p = 0.519, Fisher Exact; Clopper and Pearson exact approach

6. Secondary Outcome: Percentage of Participants Achieving an Increase From Baseline Hemoglobin of ≥2 g/dL and/or Hemoglobin ≥ 11 g/dL
Description: Percentage of participants achieving an increase from baseline hemoglobin of ≥ 2 g/dL and/or hemoglobin ≥ 11 g/dL for 28 consecutive days during the treatment period and up to 2 months after the last dose of study treatment in the absence of RBC transfusion or treatment with an ESA. The percentage of participants achieving an increase from baseline hemoglobin of ≥ 2 g/dL and/or hemoglobin ≥ 11 g/dL for 28 consecutive days is presented.
Time Frame: Baseline and Up to ~145 Days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo | All Sotatercept-treated Participants
Number analyzed (Participants) | 5 | 9 | 4 | 5 | 18
Percentage of Participants
  Overall | 20.0 [0.5 to 71.6] | 22.2 [2.8 to 60.0] | 75.0 [19.4 to 99.4] | 20.0 [0.5 to 71.6] | 33.3 [13.3 to 59.0]
  Received weekly chemotherapy and showed a response: number analyzed (Participants) | 2 | 2 | 1 | 1 | 5
  Received weekly chemotherapy and showed a response | 0 [0 to 84.2] | 11.1 [1.3 to 98.7] | 25.0 [2.5 to 100.0] | 20.0 [2.5 to 100.0] | 11.1 [5.3 to 85.3]
  Received less frequent chemotherapy and showed a response: number analyzed (Participants) | 3 | 7 | 3 | 4 | 13
  Received less frequent chemotherapy and showed a response | 20.0 [0.8 to 90.6] | 11.1 [0.4 to 57.9] | 50.0 [9.4 to 99.2] | 0 [0 to 60.2] | 22.2 [9.1 to 61.4]
Statistical Analysis 1: Comparison: Sotatercept 0.1 mg/kg vs Placebo; Overall; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 2: Comparison: Sotatercept 0.3 mg/kg vs Placebo; Overall; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 3: Comparison: Sotatercept 0.5 mg/kg vs Placebo; Overall; Test type: Superiority; p = 0.206, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 4: Comparison: Placebo vs All Sotatercept-treated Participants; Overall; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 5: Comparison: Sotatercept 0.1 mg/kg vs Placebo; Weekly Chemotherapy; Test type: Superiority; p = 0.333, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 6: Comparison: Sotatercept 0.3 mg/kg vs Placebo; Weekly Chemotherapy; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 7: Comparison: Placebo vs All Sotatercept-treated Participants; Weekly Chemotherapy; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 8: Comparison: Sotatercept 0.1 mg/kg vs Placebo; Less Frequent Chemotherapy; Test type: Superiority; p = 0.429, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 9: Comparison: Sotatercept 0.3 mg/kg vs Placebo; Less Frequent Chemotherapy; Test type: Superiority; p > 0.999, Fisher Exact — P-values greater than 0.999 are reported as ">0.999"; Clopper and Pearson exact approach
Statistical Analysis 10: Comparison: Sotatercept 0.5 mg/kg vs Placebo; Less Frequent Chemotherapy; Test type: Superiority; p = 0.143, Fisher Exact; Clopper and Pearson exact approach
Statistical Analysis 11: Comparison: Placebo vs All Sotatercept-treated Participants; Less Frequent Chemotherapy; Test type: Superiority; p = 0.519, Fisher Exact; Clopper and Pearson exact approach

7. Secondary Outcome: Duration of Hematopoietic Response for Hemoglobin ≥ 1 g/dL
Description: Duration of hematopoietic response is defined as the time period from the first time hemoglobin increases at least ≥ 1 g/dL from baseline to the last time there is hemoglobin ≥ 1 g/dL increase from baseline. Duration of response is only calculated for a responder and will be at least 28 days. The duration of response is only calculated for a patient who meets the primary efficacy endpoint. The data for duration of response for ≥ 1 g/dL from baseline is presented.
Time Frame: Baseline and Up to ~145 Days
Population: All randomized participants who have confirmed CIA, received at least one dose of study intervention, on study intervention for at least 2 months (57 days) and had a hematopoietic response of ≥1 g/dL and less than 2 g/dL increase from baseline.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 0 | 3 | 2 | 1
Days |  | 47.0 (20.30) | 46.5 (14.85) | 29.0 (NA) — NA = Standard deviation cannot be calculated for 1 participant.

8. Secondary Outcome: Duration of Hematopoietic Response for Hemoglobin ≥ 2 g/dL
Description: Duration of hematopoietic response is defined as the time period from the first time hemoglobin increases at least ≥ 2 g/dL from baseline to the last time there is hemoglobin ≥ 2 g/dL increase from baseline. Duration of response is only calculated for a responder and will be at least 28 days. The duration of response is only calculated for a patient who meets the primary efficacy endpoint. The data for duration of response for hemoglobin ≥ 2 g/dL from baseline is presented.
Time Frame: Baseline and Up to ~145 Days
Population: All randomized participants who have confirmed CIA, received at least one dose of study intervention, on study intervention for at least 2 months (57 days) and had a hematopoietic response of ≥2 g/dL and less than 11 g/dL increase from baseline.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 0 | 1 | 0 | 0
Days |  | 69.0 (NA) — NA = Standard deviation cannot be calculated for 1 participant. |  |

9. Secondary Outcome: Duration of Hematopoietic Response for Hemoglobin ≥ 11 g/dL
Description: Duration of hematopoietic response is defined as the time period from the first time hemoglobin increases at least ≥ 11 g/dL from baseline to the last time there is hemoglobin ≥ 11 g/dL increase from baseline. Duration of response is only calculated for a responder and will be at least 28 days. The duration of response is only calculated for a patient who meets the primary efficacy endpoint. The data for duration of response for hemoglobin ≥ 11 g/dL from baseline is presented.
Time Frame: Baseline and Up to ~145 Days
Population: All randomized participants who have confirmed CIA, received at least one dose of study intervention, on study intervention for at least 2 months (57 days), and had a hematopoietic response of ≥11 g/dL increase from baseline.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 0 | 1 | 2 | 1
Days |  | 41.0 (NA) — NA = Standard deviation cannot be calculated for 1 participant. | 50.0 (9.90) | 29.0 (NA) — NA = Standard deviation cannot be calculated for 1 participant.

10. Secondary Outcome: Duration of Hematopoietic Response for Hemoglobin Increases ≥ 1 g/dL and/or Hemoglobin Concentration ≥ 11 g/dL
Description: Duration of hematopoietic response is defined as the time period the first time hemoglobin increases ≥ 1 g/dL and/or hemoglobin concentration is ≥ 11 g/dL from baseline to the last time when the same response is maintained. The data for duration of response for hemoglobin ≥ 1 g/dL and/or hemoglobin concentration ≥ 11 g/dL from baseline is presented.
Time Frame: Baseline and Up to ~145 Days
Population: All randomized participants who have confirmed CIA, received at least one dose of study intervention, on study intervention for at least 2 months (57 days), and had a hematopoietic response of ≥ 1 g/dL and/or hemoglobin concentration is ≥11 g/dL increase from baseline.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 0 | 3 | 2 | 1
Days |  | 47.0 (20.30) | 50.0 (9.90) | 29.0 (NA) — NA = Standard deviation cannot be calculated for 1 participant.

11. Secondary Outcome: Duration of Hematopoietic Response for Hemoglobin Increases ≥ 2 g/dL, and/or Hemoglobin Concentration ≥ 11 g/dL
Description: Duration of hematopoietic response is defined as the time period the first time hemoglobin increases ≥ 2 g/dL, and/or hemoglobin concentration is ≥ 11 g/dL from baseline to the last time when the same response is maintained. The data for duration of response for hemoglobin ≥ 2 g/dL and/or hemoglobin concentration ≥ 11 g/dL from baseline is presented.
Time Frame: Baseline and Up to ~145 Days
Population: All randomized participants who have confirmed CIA, received at least one dose of study intervention, on study intervention for at least 2 months (57 days) and had a hematopoietic response of ≥ 2 g/dL and/or hemoglobin concentration is ≥11 g/dL increase from baseline.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 0 | 1 | 2 | 1
Days |  | 69.0 (NA) — NA = Standard deviation cannot be calculated for 1 participant. | 50.0 (9.90) | 29.0 (NA) — NA = Standard deviation cannot be calculated for 1 participant.

12. Secondary Outcome: Time to Achieve Hematopoietic Response of Hemoglobin ≥ 1 g/dL Increase From Baseline
Description: Time to achieve hematopoietic response based on ≥ 1 g/dL increase from baseline, is defined as the time from first dose of study treatment to the first hemoglobin increase ≥ 1 g/dL that was maintained for at least 28 consecutive days. The data for time to achieve hematopoietic response for hemoglobin ≥ 1 g/dL from baseline is presented.
Time Frame: Baseline and Up to ~145 Days
Population: All randomized participants who have confirmed CIA, received at least one dose of study intervention, on study intervention for at least 2 months (57 days) and had a hematopoietic response of ≥ 1 g/dL increase from baseline.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 0 | 3 | 2 | 1
Days |  | NA [72.0 to NA] — NA = Not estimable due to small number of responses. | NA [6.0 to NA] — NA = Not estimable due to small number of responses. | NA [112 to NA] — NA = Not estimable due to small number of responses.

13. Secondary Outcome: Time to Achieve Hematopoietic Response of Hemoglobin ≥ 2 g/dL Increase From Baseline
Description: Time to achieve hematopoietic response based on ≥ 2 g/dL increase from baseline, is defined as the time from first dose of study treatment to the first hemoglobin increase ≥ 2 g/dL that was maintained for at least 28 consecutive days. The data for duration of response for hemoglobin ≥ 2 g/dL from baseline is presented.
Time Frame: Baseline and Up to ~145 Days
Population: All randomized participants who have confirmed CIA, received at least one dose of study intervention, on study intervention for at least 2 months (57 days) and had a hematopoietic response of ≥ 2 g/dL increase from baseline.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 0 | 1 | 0 | 0
Days |  | NA [NA to NA] — NA = Not estimable due to small number of responses. |  |

14. Secondary Outcome: Time to Achieve Hematopoietic Response of Hemoglobin ≥ 11 g/dL From Baseline
Description: Time to achieve hematopoietic response based on hemoglobin ≥ 11 g/dL, defined as the time from first dose of study treatment to the first hemoglobin ≥ 11 g/dL that was maintained for at least 28 consecutive days. The data for duration of response for hemoglobin ≥ 11 g/dL from baseline is presented.
Time Frame: Baseline and Up to ~145 Days
Population: All randomized participants who have confirmed CIA, received at least one dose of study intervention, on study intervention for at least 2 months (57 days) and had hematopoietic response of ≥ 11 g/dL increase from baseline.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 1 | 2 | 3 | 1
Days | NA [28.0 to NA] — NA = Not estimable due to small number of responses. | NA [100.0 to NA] — NA = Not estimable due to small number of responses. | 56.0 [6.0 to NA] — NA = Not estimable due to small number of responses. | NA [112.0 to NA] — NA = Not estimable due to small number of responses.

15. Secondary Outcome: Time to Achieve Hematopoietic Response of First Hemoglobin Increase ≥ 1 g/dL and/or Hemoglobin ≥ 11 g/dL
Description: Time to achieve hematopoietic response based on multiple criteria categories, defined as the time from first dose of study treatment to first hemoglobin increase ≥ 1 g/dL and/or hemoglobin ≥ 11 g/dL that was maintained for at least 28 consecutive days. The data for duration of response for hemoglobin increase from baseline ≥ 1 g/dL and/or ≥ 11 g/dL from baseline is presented.
Time Frame: Baseline and Up to ~145 Days
Population: All randomized participants who have confirmed CIA, received at least one dose of study intervention, on study intervention for at least 2 months (57 days) and had a hematopoietic response of ≥ 1 g/dL and/or hemoglobin concentration is ≥11 g/dL increase from baseline.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 1 | 4 | 3 | 1
Days | NA [28.0 to NA] — NA = Not estimable due to small number of responses. | NA [21.0 to NA] — NA = Not estimable due to small number of responses. | 56.0 [6.0 to NA] — NA = Not estimable due to small number of responses. | NA [112.0 to NA] — NA = Not estimable due to small number of responses.

16. Secondary Outcome: Time to Achieve Hematopoietic Response of First Hemoglobin Increase ≥ 2 g/dL and/or Hemoglobin ≥ 11 g/dL
Description: Time to achieve hematopoietic response, defined as the time from first dose of study treatment to first hemoglobin increase ≥ 2 g/dL and/or hemoglobin ≥ 11 g/dL that was maintained for at least 28 consecutive days. The data for duration of response for hemoglobin increase from baseline ≥ 2 g/dL and/or ≥ 11 g/dL from baseline is presented.
Time Frame: Baseline and Up to ~145 Days
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 1 | 2 | 3 | 1
Days | NA [28.0 to NA] — NA = Not estimable due to small number of responses. | NA [NA to NA] — NA = Not estimable due to small number of responses. | 56.0 [6.0 to NA] — NA = Not estimable due to small number of responses. | NA [112.0 to NA] — NA = Not estimable due to small number of responses.

17. Secondary Outcome: Percentage of Participants Who Received RBC Transfusion or Treatment With an ESA
Description: The percentage of participants who received RBC transfusion or treatment with an ESA in each study treatment group as well as within each cycle of each study treatment is presented.
Time Frame: Up to Day 141
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 5 | 9 | 4 | 5
Percentage of Participants
  Overall RBC Transfusions | 0 | 33.3 | 25.0 | 0
  Overall ESAs | 0 | 11.1 | 0 | 0
  Overall Received RBC Transfusions or ESAs | 0 | 44.4 | 25.0 | 0
  Day 1 to Prior to Day 29 RBC Transfusions | 0 | 11.1 | 25.0 | 0
  Day 1 to Prior to Day 29 ESAs | 0 | 0 | 0 | 0
  Day 1 to Prior to Day 29 Received RBC Transfusions or ESAs | 0 | 11.1 | 25.0 | 0
  Day 29 to Prior to Day 57 RBC Transfusions | 0 | 22.2 | 0 | 0
  Day 29 to Prior to Day 57 ESAs | 0 | 0 | 0 | 0
  Day 29 to Prior to Day 57 Received RBC Transfusions or ESAs | 0 | 22.2 | 0 | 0
  Day 57 to Prior to Day 85 RBC Transfusions | 0 | 0 | 25.0 | 0
  Day 57 to Prior to Day 85 ESAs | 0 | 11.1 | 0 | 0
  Day 57 to Prior to Day 85 Received RBC Transfusions or ESAs | 0 | 11.1 | 25.0 | 0
  Day 85 to Prior to Day 141 RBC Transfusions | 0 | 11.1 | 25.0 | 0
  Day 85 to Prior to Day 141 ESAs | 0 | 0 | 0 | 0
  Day 85 to Prior to Day 141 Received RBC Transfusions or ESAs | 0 | 11.1 | 25.0 | 0

18. Secondary Outcome: Objective Response Rate (ORR) for Target Lesions at Day 64 Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v 1.1).
Description: ORR is defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. The percentage of participants who experienced a CR or PR at Day 64 is presented.
Time Frame: Baseline and Day 64
Population: All randomized participants who have confirmed CIA, received at least one dose of study intervention, on study intervention for at least 2 months (57 days) and had a response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 4 | 6 | 2 | 4
Percentage of Participants
  Complete Response | 0 | 33.3 | 0 | 0
  Partial Response | 0 | 16.7 | 0 | 0
  Stable Disease | 100.0 | 16.7 | 100.0 | 50.0
  Progressive Disease | 0 | 16.7 | 0 | 0
  Not Evaluable | 0 | 0 | 0 | 0
  Not Applicable | 0 | 16.7 | 0 | 50.0

19. Secondary Outcome: Objective Tumor Response Rate for Non-target Lesions at Day 64 Using RECIST v 1.1.
Description: ORR is defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. The percentage of participants who experienced a CR or PR of non-target lesions at Day 64 is presented.
Time Frame: Day 64
Population: as for outcome 18
Measure: Number; unit: Percentage of Participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 4 | 6 | 2 | 4
Percentage of Participants
  Complete Response | 0 | 0 | 0 | 0
  Progressive Disease | 50.0 | 33.3 | 0 | 50.0
  Non-complete Response/Non-progressive disease | 50.0 | 50.0 | 100.0 | 25.0
  Not Evaluable | 0 | 0 | 0 | 0
  Not Applicable | 0 | 16.7 | 0 | 25.0

20. Secondary Outcome: Objective Tumor Response Rate for Target Lesions on Day 113 Using RECIST v 1.1.
Description: ORR is defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. The percentage of participants who experienced a CR or PR at Day 113 is presented.
Time Frame: Day 113
Population: as for outcome 18
Measure: Number; unit: Percentage of Participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 3
Percentage of Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0
  Stable Disease | 100.0 | 0 | 0 | 33.3
  Progressive Disease | 0 | 0 | 0 | 0
  Not Evaluable | 0 | 0 | 0 | 0
  Not Applicable | 0 | 100.0 | 100.0 | 66.7

21. Secondary Outcome: Objective Tumor Response Rate for Non-target Lesions on Day 113 Using RECIST v 1.1.
Description: ORR is defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. The percentage of participants who experienced a CR or PR of non-target lesions at Day 113 is presented.
Time Frame: Day 113
Population: as for outcome 18
Measure: Number; unit: Percentage of Participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo
Number analyzed (Participants) | 2 | 2 | 1 | 3
Percentage of Participants
  Complete Response | 0 | 0 | 0 | 0
  Progressive Disease | 0 | 0 | 100.0 | 33.3
  Non-complete Response/Non-progressive disease | 100.0 | 50.0 | 0 | 33.3
  Not Evaluable | 0 | 50.0 | 0 | 0
  Not Applicable | 0 | 0 | 0 | 33.3

22. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from start of the chemotherapy regimen (which could have occurred prior to study start and collected as prior anticancer therapy) to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS per RECIST 1.1 is presented.
Time Frame: From start of chemotherapy (which could have occurred prior to study start) up to Study Day 281
Population: All randomized participants who received at least one dose of study intervention.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo | All Sotatercept-treated Participants
Number analyzed (Participants) | 8 | 10 | 7 | 5 | 25
Days | 188.0 [64.0 to 188.0] | 196.0 [97.0 to 219.0] | 187.0 [134.0 to 1791.0] | 157.0 [84.0 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 169.0 [108.0 to 219.0]

ADVERSE EVENTS:
Time Frame: Up to Day 281
Description: The safety analysis population included all participants who received at least one dose of study treatment. The analysis population for All-Cause Mortality included all allocated participants.
Groups:
- Total: Total for all participants
Arm/Group | Sotatercept 0.1 mg/kg | Sotatercept 0.3 mg/kg | Sotatercept 0.5 mg/kg | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 1/8 | 3/10 | 3/7 | 0/5 | 7/30
Serious Adverse Events (participants affected / at risk) | 0/8 | 2/10 | 3/7 | 1/5 | 6/30
Other Adverse Events (participants affected / at risk) | 6/8 | 7/10 | 7/7 | 5/5 | 25/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept 0.1 mg/kg (N=8) | Sotatercept 0.3 mg/kg (N=10) | Sotatercept 0.5 mg/kg (N=7) | Placebo (N=5) | Total (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotatercept 0.1 mg/kg (N=8) | Sotatercept 0.3 mg/kg (N=10) | Sotatercept 0.5 mg/kg (N=7) | Placebo (N=5) | Total (N=30)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 7 (7)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (8) | 0 (0) | 0 (0) | 2 (4) | 5 (12)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 4 (9) | 0 (0) | 2 (3) | 3 (7) | 9 (19)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 1 (6) | 0 (0) | 4 (10)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (5) | 3 (5) | 6 (12)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peritoneal effusion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 5 (6)
Asthenia (General disorders) | 3 (3) | 2 (2) | 2 (4) | 2 (3) | 9 (12)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 6 (6)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Device migration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin turgor decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal identification test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5) | 2 (2) | 0 (0) | 4 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metastases to gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (5) | 5 (8)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Enuresis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
This is an acquired study. No restrictions were imposed on time on current chemotherapy prior to study entry, therefore PFS could have gone beyond the study duration. The time from start of current chemotherapy could have occurred prior to study start and collected as prior anticancer therapy, therefore the upper limit of the confidence interval in the "Sotatercept 0.5 mg/kg" arm, "1791.0 days", didn't exceed the timeframe of 281 days after study start.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information concerning Sotatercept is considered confidential and shall remain the sole property of the Sponsor. No publication or disclosure of study results will be permitted except as specified in a separate, written, agreement between the Sponsor and the Investigator.

DOCUMENTS (2):
  • Study Protocol (2009-03-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT00931606/Prot_000.pdf
  • Statistical Analysis Plan (2009-10-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT00931606/SAP_001.pdf